CLINICAL TRIAL: NCT05661162
Title: Evaluation of the Effect of the "CR500 SINGLE-DOSE GEL" Medical Device in Patients With Knee Osteoarthritis (KOA): a Post-market Confirmatory Interventional, Single Arm Clinical Investigation
Brief Title: Evaluation of the Effect of the "CR500 SINGLE-DOSE GEL" Medical Device in Patients With Knee Osteoarthritis (KOA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contrad Swiss SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTD-SW CR500-KOA 2020
Record Dates: First submitted 2022-11-16; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis;; Hyaluronic acid; Peptides; Synovial fluid; Algofunctional scores; Biochemical markers; Macrophages infiltration
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CR500 single-dose gel (Other): Interventional study on CR500 1.5 mL will be topically administered twice a week for four weeks
  Interventions: Device: CR 500™ SINGLE-DOSE GEL

INTERVENTIONS:
Device: CR 500™ SINGLE-DOSE GEL — CR 500™ SINGLE-DOSE GEL is a hydrogel to be applied to intact skin, useful to attenuate the physiological degeneration of cartilage typical of osteoarthritic processes. The presence of sodium hyaluronate facilitates the movement of joints and tendons for greater mobility and flexibility

SUMMARY:
Single arm clinical investigation, post-market confirmatory interventional to assess performance, safety and tolerability of "CR500 SINGLE-DOSE GEL" medical device in patients with knee osteoarthritis (KOA).

DETAILED DESCRIPTION:
Subjects 26-83 years old will receive CR500 SINGLE-DOSE GEL given for the treatment of osteoarthritis of the knee over a 4-week time period. The primary objective of the study is to evaluate the effect of CR500 SINGLE-DOSE GEL in the treatment of KOA.

ELIGIBILITY:
Inclusion criteria

1. Male or Female, aged ≥18 years at the time of the signature of ICF (Informed Consent Form).
2. Patients with a diagnosis of primary or secondary KOA affecting only one knee (monolateral KOA) of "mild" (score 1 - 4) or "moderate" (score 5 - 7) severity according to the LKI score.
3. Willing to follow all study procedures, including attending all site visits, tests and examinations.
4. Willing to participate in the study and sign the ICF.

Exclusion criteria

1. Osteoarthritis (OA) in both knees (bilateral KOA).
2. Other - different - clinical conditions of the knee.
3. Infective or inflammatory processes near the area of treatment.
4. Damaged skin in the area of treatment.
5. Ongoing cutaneous allergies.
6. Serious and chronical pathological skin conditions (i.e. rosacea, psoriasis, vitiligo) including diagnosticated cancer with/without ongoing antitumor therapy.
7. Allergy to device components (Sodium hyaluronate; Synthetic Human (SH)-Polypeptide-85; SH-Polypeptide-93; Glycerin; Propylene glycol; Ethylhexylglycerin; Panthenol; Polyethylene Glycol (PEG)-40 hydrogenated castor oil; Sodium hydroxide; Xanthan gum; Phenoxyethanol; Benzoic Acid; Carbomer; Dehydroacetic Acid; Disodium EDTA).
8. Any other systemic or local therapy for the treatment of KOA.
9. Any other systemic or local therapy (e.g. NSAIDs, corticosteroids) for the treatment of other inflammatory diseases (e.g. dermatitis, acute or chronic bronchitis, gastroenteritis, etc.) or painful states (e.g. headache, dental abscess, etc.) that may interfere with the clinical course of KOA under treatment with the medical device CR500.
10. Immune system illnesses.
11. Uncontrolled systemic diseases.
12. Known drug and/or alcohol abuse.
13. Mental incapacity that precludes adequate understanding or cooperation.
14. Participation in another investigational study.
15. Pregnancy* or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
OA evaluation, measured by Lequesne Knee Index (LKI) | 4 weeks
  The primary efficacy endpoint of the study will be the evaluation of the clinical performance of the CR 500™, used as intended in patients affected by KOA, in variation of symptoms related to the physiological degeneration of cartilage typical of osteoarthritic processes, in terms of difference in LKI score between the end study visit and baseline visit.
  Lequesne Knee Index Score:
  minimum index score: 0 maximum index score: 24
  0 means none OA
  >= means extremely severe OA

SECONDARY OUTCOMES:
Lequesne Knee Index (LKI) Score | 4 weeks
  To evaluate the clinical performance of the CR 500™ across the study by Lequesne Knee Index (LKI) score.
  Lequesne Knee Index Score:
  minimum index score: 0 maximum index score: 24
  0 means none OA
  >= means extremely severe OA
Lequesne Knee Index (LKI) Subscore | 4 weeks
  To evaluate the clinical performance of the CR 500™ by each Lequesne Knee Index (LKI) subscore
  Lequesne Knee Index Score:
  minimum index score: 0 maximum index score: 24
  0 means none OA
  >= means extremely severe OA
Symptoms Variation in terms of Lequesne Knee Index (LKI) score | 4 weeks
  To evaluate the clinical performance of the CR 500™ in the attenuation of symptoms in patients affected by KOA stratified by KOA severity as assessed by Lequesne Knee Index (LKI) score
Cluster of Subjective Symptoms evaluated by Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire | 4 weeks
  To evaluate the different dimensions of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
  Koos converted into a 0-100 Score
  0 means worst level of OA 100 means best level of OA
  Subscores:
  Pain, Symptoms, Sports, Quality of Life, Activities of Daily Living
Number of participants with treatment-related adverse event as assessed by a questionnaire. | 4 weeks
  To evaluate the side effects of the product CR 500™ through a the completion of a specific questionnaire by the patient.
Product tolerability and patient satisfaction as assessed by a questionnaire using a five-points Likert scale | 4 weeks
  To evaluate the tolerability and patient satisfaction of the CR 500™ through a the completion of a specific questionnaire by the patient, the five-points Likert scale in which 1 means Strongly disagree with the assertion and 5 means Strongly agree
Evaluation of the status of the cartilage degradation by quantification of neoepitope of type II collagen (C2C) | 4 weeks
  Evaluation of the status of the cartilage degradation by quantification of neoepitope of type II collagen in synovial fluid by ELISA (ng/mL)
Evaluation of the status of the cartilage degradation by quantification of C-terminal telopeptide of type II collagen (CTX-II) | 4 weeks
  Evaluation of the status of the cartilage degradation by quantification of C-terminal telopeptide of type II collagen quantification (CTX-II) in synovial fluid by ELISA (pg/mL)
Evaluation of the status of the cartilage by quantification of type II collagen propeptide (CPII) quantification | 4 weeks
  Evaluation of the status of the cartilage by quantification of type II collagen propeptide (CPII) in synovial fluid by ELISA (ng/mL)
Evaluation of the status of the cartilage by quantification of hyaluronic acid (HA) quantification | 4 weeks
  Evaluation of the status of the cartilage by quantification of hyaluronic acid (HA) in synovial fluid by ELISA (mg/mL)
Evaluation of the inflammatory status of the knee joint by quantification of tumour necrosis factor (TNF) quantification | 4 weeks
  Evaluation of the status of the cartilage by quantification of tumour necrosis factor (TNF) in synovial fluid by ELISA (pg/mL)
Evaluation of the macrophages infiltration in the knee joint by quantification of Cluster of Differentiation 206 (CD206) | 4 weeks
  Evaluation of the macrophages infiltration in the knee joint by quantification of Cluster of Differentiation 206 (CD206) by Real Time Polymerase Chain Reaction (PCR)
Evaluation of the macrophages infiltration in the knee joint by quantification of Cluster of Differentiation 11c (CD11c) | 4 weeks
  Evaluation of the macrophages infiltration in the knee joint by quantification of Cluster of Differentiation 11c (CD11c) by Real Time PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Mater Domini Casa di Cura Privata - Gruppo Humanitas, Castellanza, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Colombini A, Doro G, Ragni E, Forte L, de Girolamo L, Zerbinati F. Treatment with CR500(R) improves algofunctional scores in patients with knee osteoarthritis: a post-market confirmatory interventional, single arm clinical investigation. BMC Musculoskelet Disord. 2023 Aug 12;24(1):647. doi: 10.1186/s12891-023-06754-7. PMID 37573322